CLINICAL TRIAL: NCT01096537
Title: Evolution of the Incidence of Occupational Asthma at the Beginning of the Activity of Young Bakers, Pastry-makers and Hairdressers, and Exploration of Its Risk Factors
Brief Title: Early Incidence of Occupational Asthma Among Bakers, Pastry-makers and Hairdressers
Acronym: ABCD
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University of Nancy (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-A00622-53
Record Dates: First submitted 2010-03-10; First posted 2010-03-31 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-03

CONDITIONS: Occupational Asthma
Keywords: incidence; young workers; occupations at risk; public health; epidemiology; polymorphisms; gentic
MeSH Terms: conditions — Asthma, Occupational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Young workers: Exposed young workers graduated in sectors at risk of occupational asthma (bakery, pastry-making or hairdressing)
  "Non-exposed" young workers graduated in sectors without specific occupational exposure as the sale or the food sectors.

SUMMARY:
Background: Occupational exposures are thought to be responsible for 10-15% of new-onset asthma cases in adults, with disparities across sectors. Because most of the data are derived from registries and cross-sectional studies, little is known about incidence of occupational asthma (OA) during the first years after inception of exposure. This study focuses on this early asthma onset period among young workers in the bakery, pastry making and hairdressing sectors in order to assess early incidence of OA in these "at risk" occupations according to exposure duration, and to identify risk factors of OA.

Methods: This study is a longitudinal retrospective study with a nested case-control to identify risk factors of OA. The assessment of incidence evolution is made by exploring a series of promotions (or retrospective cohorts) with increasing duration since at work. The study population is composed of subjects who graduated between 2001 and 2006 in sectors where they experience exposure to organic or inorganic allergenic or irritant compounds (with an objective of 150 subjects by year) and 250 young workers with no specific occupational exposure.

This study is a descriptive, monocentric, longitudinal and retrospective study with cross-sectional measurements.

ELIGIBILITY:
Inclusion Criteria:

* for the exposed group: to be graduated between 2001 and 2006 from nine vocational schools in Lorraine, North-Eastern France
* for the "non-exposed" group: to be graduated in 2001 in the sale or the food sectors (butcher, pork butcher, caterer, cook job,…) from the same vocational schools

Exclusion Criteria:

* asthma diagnosed before apprenticeship
* for the "non-exposed" group: to have worked previously or later in a sector at risk with OA

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All bakers, pastry-makers and hairdressers who graduated between 2001 and 2006 from nine vocational schools in Lorraine, North-Eastern France, and all subjects who graduated in 2001 in the sale or the food sectors (butcher, pork butcher, caterer, cook job,…) from the same vocational schools.
Sampling Method: Non-Probability Sample
Enrollment: 866 (Actual)
Dates: Start 2008-12; Primary Completion 2010-01 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
The early incidence of OA among young workers according to their sector of activity and exposure duration. | 3-6 months after tle last inclusion

SECONDARY OUTCOMES:
The identification of risk factors of OA. | 3-6 months after the last inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PARIS, MD / PhD, Principal Investigator — CHU Nancy, INSERM, Nancy University; Denis ZMIROU-NAVIER, MD / PhD, Principal Investigator — INSERM, Nancy university, EHESP School of Public Health
Locations (1):
- CHU Nancy, Nancy, France

REFERENCES:
- [Derived] Remen T, Coevoet V, Acouetey DS, Gueant JL, Gueant-Rodriguez RM, Paris C, Zmirou-Navier D. Early incidence of occupational asthma among young bakers, pastry-makers and hairdressers: design of a retrospective cohort study. BMC Public Health. 2010 Apr 26;10:206. doi: 10.1186/1471-2458-10-206. PMID 20420675